CLINICAL TRIAL: NCT05079919
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of ISIS 678354 Administered Subcutaneously to Patients With Severe Hypertriglyceridemia
Brief Title: A Study of Olezarsen (ISIS 678354) Administered to Participants With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 678354-CS5; 2021-002192-19 (EudraCT Number); 2024-510696-38-00 (EU CTIS Number)
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Severe Hypertriglyceridemia
Keywords: ISIS 678354; Fasting Triglycerides; Apolipoprotein C-III; Very Low-Density Lipoprotein Cholesterol; High-Density Lipoprotein-Cholesterol; Non-High-Density Lipoprotein-Cholesterol; Olezarsen
MeSH Terms: conditions — Hypertriglyceridemia | interventions — olezarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olezarsen (Experimental): Olezarsen will be administered once every 4 weeks by subcutaneous (SC) injection from Week 1 through Week 49.
  Interventions: Drug: Olezarsen
- Placebo (Placebo Comparator): Olezarsen-matching placebo will be administered once every 4 weeks by SC injection from Week 1 through Week 49.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olezarsen — Olezarsen will be administered by SC injection.
  Other Names: AKCEA-APOCIII-LRx; ISIS 678354
  Arms: Olezarsen
Drug: Placebo — Olezarsen-matching placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of olezarsen as compared to placebo on the percent change in fasting triglycerides (TG) from baseline.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study in 617 participants. Participants will be randomized to receive olezarsen or placebo in a 53-week treatment period. The length of participation in the study will be approximately 78 weeks, which includes an up to 12-week screening period, a 53-week treatment period, and a 13-week post-treatment evaluation period or transition to open-label extension (OLE) study with up to 1-year treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Fasting TG ≥ 500 mg/dL (5.65 mmol/L) at Screening and Qualification
* Patients must be on lipid-lowering therapy that should adhere to standard of care (SOC) per local guidelines. Lipid-lowering medications should be optimized and stabilized for at least 4 weeks prior to Screening to minimize changes in these medications during the study.

Key Exclusion Criteria:

* Hemoglobin A1c (HbA1c) ≥ 9.5% at Screening
* Alanine aminotransferase or aspartate aminotransferase > 3.0 × upper limit of normal
* Total bilirubin > upper limit of normal unless due to Gilbert's syndrome
* Estimated GFR < 30 mL/min/1.73 m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Fasting TG Compared to Placebo | Baseline and Month 6

SECONDARY OUTCOMES:
Percent Change from Baseline in Fasting TG Compared to Placebo | Baseline and Month 12
Percent Change from Baseline in Fasting Apolipoprotein C-III (ApoC-III), Remnant Cholesterol and Fasting Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) Compared to Placebo | Baseline, Month 6 and 12
Proportion of Patients Who Achieve Fasting TG <500 mg/dL (5.65 mmol/L) Compared to Placebo | Month 12
Proportion of Participants Who Achieve Fasting TG < 880 mg/dL (10 mmol/L) Compared to Placebo in the Subgroup of Participants with Baseline TG ≥ 880 mg/dL | Month 12
Adjudicated Acute Pancreatitis Event Rate During the Treatment Period Compared to Placebo | Week 1 through Week 53
Absolute Change in Hepatic Fat Fraction (HFF) Between Olezarsen Treatment Group and Pooled Placebo | Baseline through Month 12

CONTACTS AND LOCATIONS:
Locations (209):
- United States (56):
  - Accel Research Sites Network, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Velocity Clinical Research, Chula Vista, California
  - Diabetes/Lipid Management & Research Center, Huntington Beach, California
  - University of California, San Diego (UCSD), La Jolla, California
  - LA Universal Research Center, Inc., Los Angeles, California
  - America Clinical Trials, Tarzana, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Southeast Clinical Research LLC, Chiefland, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Finlay Medical Research, Miami, Florida
  - Innovia Research Center, INC, Miramar, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - IMA Clinical Research, St. Petersburg, Florida
  - VICIS Clinical Research, Tampa, Florida
  - Bayside Clinical Research, Trinity, Florida
  - IACT Health, Columbus, Georgia
  - IMA Clinical Research Chicago, Chicago, Illinois
  - Affinity Health, Oak Brook, Illinois
  - West Broadway Clinic, Council Bluffs, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Clinical Trials of America, LLC, Monroe, Louisiana
  - Continental Clinical Solutions, Towson, Maryland
  - University of Michigan Hospital and Health Systems/ Dept. of Pharmacy-Research Pharmacy, Ann Arbor, Michigan
  - Aa Mrc, Llc, Flint, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - IMA Clinical Research, St Louis, Missouri
  - Bryan Medical Center Clinical Research, Lincoln, Nebraska
  - Palm Research Center, INC., Las Vegas, Nevada
  - Hudson County Clinical Trials Research Center, Union City, New Jersey
  - Modern Medicine, Brooklyn, New York
  - Northwell Health, Great Neck, New York
  - Circuit Clinical (Crystal Run Healthcare), Middletown, New York
  - NYU Langone, New York, New York
  - Columbia University, New York, New York
  - Circuit Clinical, Niagara Falls, New York
  - Modern Medical, Syosset, New York
  - Novant Health Cancer Institute Elizabeth Investigational Drug Services, Charlotte, North Carolina
  - Cone Medical Center, Greensboro, North Carolina
  - Clinical Trials of America, LLC, Mount Airy, North Carolina
  - Wake Forest University Health Sciences, Salem, North Carolina
  - Aventiv Research, Columbus, Ohio
  - Summit Research Group, LLC, Munroe Falls, Ohio
  - Hightower Clinical Trial Services, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Medford, Oregon
  - The Miriam Hospital, Providence, Rhode Island
  - Health Concepts, Rapid City, South Dakota
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - Velocity Clinical Research, Cedar Park, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Medicus Alliance Clinical Research, Sugar Land, Texas
  - Velocity Clinical, West Jordan, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - West Virginia University Heart and Vascular Institute, Morgantown, West Virginia
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shoe Hospital, Saint Leonards, New South Wales
  - Dr. Heart Pty Ltd at Cholesterol Care Australia, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton S., Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Adelaide Hospital, Adelaide
- Bulgaria (17):
  - MHAT Blagoevgrad AD, Blagoevgrad
  - Medical Center Doctor Staykov EOOD, Burgas
  - Medical Center Diamedical 2013 OOD, Dimitrovgrad
  - MHAT "Dr. Tota Venkova" AD, Gabrovo
  - Medical Center "Hera" EOOD, Montana
  - SHAT "Special Medic" Ltd, Plovdiv
  - Medical Center Rusemed EOOD, Rousse
  - DCC 1 Sliven, Sliven
  - Gabriela Zhelyazkova, Sliven
  - Medical Center Smolyan Clinical Research OOD, Smolyan
  - Medical Center Endomedical EOOD, Sofia
  - Medical Centar "KALIMAT", Sofia
  - MC Doctor Kalchev OOD, Sofia
  - UMHAT Sofiamed OOD, Sofia
  - New Rehabilitation Center, Stara Zagora
  - UMHAT Prof. Dr. Stoyan Kirkovich AD, Clinic of Cardiology, Stara Zagora
  - Medical Centre Nevromedics EOOD, Veliko Tarnovo
- Canada (5):
  - Arc Biosystems, Vancouver, British Columbia
  - Canadian Phase Onward Inc, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Institut de recherches cliniques de Montréal (IRCM), Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
- Czechia (8):
  - MEDICUS SERVICES s.r.o., Brandýs nad Labem
  - EDUMED s.r.o., Hradec Králové
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - EDUMED s.r.o., Náchod
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice, Prague
  - Lekarna Poliklinika Hurka, Prague
  - Interni Ambulance, Uherské Hradiště
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Esbjerg Hospital, Esbjerg
  - Bispebjerg Hospital, Frederiksberg
  - Herlev Hospital, Herlev
  - Godstrup Regional Hospital, Herning
  - Regionshospitalet Viborg, Viborg
- Finland (2):
  - Turku University Hospital, Turku
  - Ylitornio Health Care Center, Ylitornio
- France (6):
  - Hôpital Louis Pradel, Bron
  - CHU Dijon Bourgogne, Dijon
  - Hopital de la Conception, Marseille
  - CHU Montpellier - Hôpital Lapeyronie, Montpellier
  - Hopital Pitie Salpetriere APHP, Paris
  - CHU Nantes - Hopital Nord Laennec, Saint-Herblain
- Germany (9):
  - Stoffwechselcentrum Charite Campus Virchow, Berlin
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - St. Josefskrankenhaus,, Heidelberg
  - Praxis Dr. med. Taggeselle, Markkleeberg
  - Kardiologische Praxis in Papenburg, Papenburg
  - Evangelisches Krankenhaus Witten, Witten
- Hungary (11):
  - BKS Research Kft, Hatvan, Heves County
  - Medifarma 98 Kft, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - CRU Hungary Kft, Borsod
  - Észak-Pesti Centrumkórház - Honvédkórház; II. Belgyógyászati Osztály, Budapest
  - Semmelweis Egyetem Kardiológiai Rehabilitacio, Budapest
  - Belinus BT, Debrecen
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszat A epulet, Debrecen
  - IPR Hungary Kft., Miskolc
  - Borbanya Praxis Eü KFT, Nyíregyháza
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - DRC Gyogyszervizsgalo Kozpont Kft, Veszprém
- Israel (9):
  - SOROKA Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Hebrew University Ein Kerm MC, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di SantOrsola, Bologna
  - Ospdale E. Bassini, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - A.O. Policlinico Universitario P. Giaccone, Palermo
  - Policlinico Umberto, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
- Netherlands (7):
  - Academic Medical Center - Department of Vascular Medicine, Amsterdam
  - Rijnstate Arnhem, Arnhem
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (3):
  - Auckland City Hospital, Grafton, Auckland
  - New Zealand Clinical Research, Christchurch
  - Wellington Regional Hospital, Newtown
- Lipid Clinic, Oslo, Norway
- Poland (6):
  - Salvia, Katowice
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - ClinMedica Research Sp.z o.o., Skierniewice
  - Osrodek Badan Klinicznych Metabolica, Tarnów
  - Futuremeds sp. z o.o, Wroclaw
  - Instytut Centrum Zdrowia Matki Polki Klinika, Łódz
- Portugal (5):
  - Centro Hospitalar do Baixo Vouga Hospital Infante D. Pedro, Aveiro
  - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Hospital Egas Moniz - Centro Hospitalar de Lisboa Ocidental, Lisbon
  - Centro Hospitalar Universitário de São João Consultas Externas de Endocrinologia K13, Porto
  - Centro Hospitalar, Vila Nova de Gaia
- Slovakia (6):
  - Medispektrum s.r.o., diabetologicka a metabolicka ambulancia, Bratislava
  - Nemocnica s poliklinikou Brezno, Brezno
  - Human-Care s.r.o., Košice
  - Vychodoslovensky Ustav srdcovych a cievnych chorob a.s., Košice
  - Cardio D&R, Košice
  - Nemocnica arm. generala L. Svobodu Svidnik,, Svidník
- South Africa (6):
  - Iatros International, Bloemfontein, Free State
  - Unitas Hospital, Centurion, Gauteng
  - Dr Jan Engelbrecht and Ass. Inc, Cape Town, Western Cape
  - TREAD Research - Department of Cardiology, Parow, Western Cape
  - University of Cape town - Lipid Factory, Cape Town
  - Chatsmed Garden Hospital, Chatsworth
- Spain (10):
  - Hospital Abente y Lago, A Coruña
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Institut d'Investigació i Innovació Parc Taulí (I3PT) Departament Medicina Universitat, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario, Madrid
  - Hospital Virgen del Rocio Edificio Centro de Diagnostico y Tratamiento (CDT), Seville
  - Hospital Universitari Sant Joan de Reus., Tarragona
- Sweden (2):
  - Sahlgrenska, University Hospital, Gothenburg, Västra Götaland County
  - Karolinska University Hospital Huddinge, Stockholm
- Turkey (Türkiye) (4):
  - Hacettepe University Medical Faculty, Ankara
  - Ege University School of Medicine, Department of Cardiology, Izmir
  - Kocaeli University Faculty of Medicine, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
- United Kingdom (16):
  - Oak Tree Surgery and Pensilva Health Centre, Liskeard, Cornwall
  - Newquay Health Centre, Newquay, Cornwall
  - Upton Surgery, Poole, Dorset
  - Panthera Biopartners, Rochdale, England
  - Panthera Biopartners, Sheffield, England
  - Huddersfield Royal Infirmary, Lindley, Huddersfield
  - Lakeside Healthcare at Corby, Corby, Northamptonshire
  - Sandwell General Hospital, Lyne, West Bromwich
  - Waterloo Medical Centre, Blackpool
  - Mounts Bay Medical Hub, Cornwell
  - Panthera, Glasgow
  - Hull Royal Infirmary, Hull
  - Panthera, London
  - Manchester University NHS Foundation Trust (MFT), Manchester
  - Panthera, Preston
  - Primary Care Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/

REFERENCES:
- [Derived] Marston NA, Bergmark BA, Alexander VJ, Prohaska TA, Kang YM, Moura FA, Zimerman A, Waldman E, Weinland J, Murphy SA, Goodrich EL, Zhang S, Xia S, Li D, Goldberg AC, Goudev A, Badimon L, Kiss RG, Vrablik M, Gaudet D, Moulin P, Stroes ESG, Banach M, Cohen H, Blom D, Charng MJ, Nordestgaard BG, Nicholls SJ, Tsimikas S, Giugliano RP, Sabatine MS; CORE-TIMI 72a and CORE2-TIMI 72b Investigators. Olezarsen for Managing Severe Hypertriglyceridemia and Pancreatitis Risk. N Engl J Med. 2026 Jan 29;394(5):429-441. doi: 10.1056/NEJMoa2512761. Epub 2025 Nov 8. PMID 41211918
- [Derived] Marston NA, Bergmark BA, Alexander VJ, Karwatowska-Prokopczuk E, Kang YM, Moura FA, Prohaska TA, Zimerman A, Zhang S, Murphy SA, Tsimikas S, Giugliano RP, Sabatine MS. Design and rationale of the CORE-TIMI 72a and CORE2-TIMI 72b trials of olezarsen in patients with severe hypertriglyceridemia. Am Heart J. 2025 Aug;286:125-135. doi: 10.1016/j.ahj.2025.03.003. Epub 2025 Mar 9. PMID 40064331